CLINICAL TRIAL: NCT00000207
Title: Multicenter Clinical Trial of Buprenorphine
Brief Title: Multicenter Clinical Trial of Buprenorphine - 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06082-3; R18DA006082 (NIH); R18-06082-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Opioid-Related Disorders
Keywords: Buprenorphine; Opioid
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to test the efficacy and safety of buprenorphine.

DETAILED DESCRIPTION:
12 different sites for a total of 736 subjects (60 at Pizarro, 70 at West LA Tx center, 15 in the 1 year extension)

ELIGIBILITY:
Inclusion Criteria:

M/F, ages 21-50. opiate dependence according to DSM-IV criteria. Self-reported use within the last 30 days. Agreeable to conditions of the study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative-hynotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1992-05; Primary Completion 1997-04 (Actual)

PRIMARY OUTCOMES:
Retention
Opiate use
Opiate craving

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States

REFERENCES:
- [Background] 1) Bup maintenance Tx of opiate dependence: A multicenter randomized tiral (Addiction, submitted) 2) Bup as a pharmacotherapy for opiate addiction: What dose provides a therapeutic response? (Am J Add 1996;5(3): 220-222.. (1) Buprenorphine maintenance treatment of opiate dependence: A multicenter randomized trial ( Addiction, submitted). (2) Buprenorphine as a pharmacotherapy for opiate addiction: What dose provides a therapeutic response? (Am J Add 1996; 5(3):220-222.